CLINICAL TRIAL: NCT02875535
Title: Implementing School Nursing Strategies to Reduce Lesbian, Gay, Bisexual, Transgender, and Queer (LGBTQ) Adolescent Suicide
Brief Title: Implementing Evidence Informed Practices in Schools to Address LGBTQ Adolescent Suicide
Acronym: RLAS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: University of New Mexico (Other); University of California, San Diego (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Cathleen Willging, Center Director, Pacific Institute for Research and Evaluation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0838.01.01; R01HD083399 (NIH)
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Suicide
Keywords: Evidence-based; lesbian, gay, bisexual, transgender, intersex, and queer; adolescent; Suicide prevention; Implementation study
MeSH Terms: conditions — Suicide; Homosexuality, Female; Homosexuality; Bisexuality; Ovotesticular Disorders of Sex Development; Suicide Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Standard school nurse care for suicide prevention.
- Dynamic Adaption Process (Experimental): Investigators will train school nurses statewide. Using the Dynamic Adaptation Process, the nurses will then convene and lead Implementation Resource Teams (IRTs). With the assistance of RLAS coaches, the school nurse-led IRTs will engage in an iterative process of assessment and planning to build school capacity and implement up to six evidence-base strategies to reduce adolescent suicide.
  Interventions: Behavioral: RLAS

INTERVENTIONS:
Behavioral: RLAS — The implementation model for this intervention will increase school-based supports and safety for gender and sexual minorities and broader student bodies, and be applicable to addressing other priority child and adolescent health and mental health issues within schools. The investigators refer to the model as "RLAS" (Implementing School Nursing Strategies to Reduce LGBTQ Adolescent Suicide).
  Other Names: Dynamic Adaptation Process
  Arms: Dynamic Adaption Process

SUMMARY:
Reducing youth suicide in the U.S. is a national public health priority. Sexual and gender minority adolescents are at elevated risk for suicide. Safer school environments, however, can decrease this risk. This study capitalizes on the critical role of school nurses in improving the mental health of this vulnerable population through implementation and sustainment of evidence-based strategies to enhance school environments. In addition to suicide, the conceptual framework and methods for this novel, nurse-led intervention can be applied to address the health-related concerns of other pediatric populations encountered in school settings as well.

DETAILED DESCRIPTION:
Reducing youth suicide in the U.S. is a national public health priority. A supportive and safe school environment is pivotal to preventing youth suicide, and schools are now widely accepted as part of the de facto mental healthcare infrastructure for adolescents. Lesbian, gay, bisexual, transgender, and queer (LGBTQ) youth are at elevated risk for suicide. Safer school environments decrease this risk. The school nurse is well positioned to implement evidence-based (EB) strategies to enhance school environments and improve the mental health of all students, particularly members of this vulnerable population. These strategies include the creation of "safe spaces," adoption of harassment and bullying prohibitions, improved access to community health and mental health providers experienced in working with youth and LGBTQ people, school staff development, and incorporation of LGBTQ-specific information into health education curricula. These strategies promote positive mental health outcomes for LGBTQ youth, and their cisgender, heterosexual peers as well.

The investigators of this nursing intervention model is called "RLAS" (Implementing School Nursing Strategies to Reduce LGBTQ Adolescent Suicide). The model builds on the Exploration, Preparation, Implementation, and Sustainment conceptual framework and the Dynamic Adaptation Process (DAP), a structured methodology for implementing the EB strategies. The DAP accounts for the multi-level context of school settings, facilitates appropriate expertise and feedback to make them "implementation ready," and provides for targeted training of school nurses. Per the DAP, the nurses and other school professionals will convene and lead Implementation Resource Teams (IRTs) consisting of counselors, social workers, health educators, and youth. With the guidance of coaches, the IRTs will engage in an iterative process of assessment and planning to build school capacity and implement the EB strategies. To evaluate this model, the investigators will combine qualitative methods with population-based surveys and pursue three specific aims.

First, the investigators will utilize the DAP to enable specially-trained nurse champions and IRTs to implement and sustain EB strategies to address the needs of LGBTQ high school students. Second, the investigators will conduct a cluster randomized controlled trial (RCT) to assess whether sexual minority students and their peers in RLAS schools report reductions in suicidality, depression, substance use, and bullying, and increased safety compared to those in usual care schools. Third, the investigators will examine the individual, school, and community factors influencing both implementation and outcomes. The RLAS keeps with national priorities to: (a) improve school-based services for pediatric populations; (b) focus on LGBTQ youth mental health; and (c) revolutionize the role of nurses in U.S. healthcare. Through its collaborative processes to refine, improve, and sustain EB strategies in these systems, the RLAS also represents a novel and innovative contribution to implementation science.

ELIGIBILITY:
Inclusion Criteria for schools:

* Located within New Mexico;
* Designated public high school;
* School nurse that is willing and available to support the RLAS intervention and to lead and convene an IRT; and
* School administrator that is willing and available to support the RLAS intervention.

Exclusion criteria for schools:

* Unable to participate in the NM-YRRS.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-05; Primary Completion 2021-12-31 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to EB strategy implementation | 5 years
  Demonstration of adherence to the Centers for Disease Control and Prevention recommended EB strategies to enhance school environments

SECONDARY OUTCOMES:
Reduced suicidality and depression measured by the New Mexico Youth Risk and Resiliency Study (NM-YRRS) | 5 years
  Self-reported suicidality and depression for youth as measured by the NM-YRRS
Substance use measured by the NM-YRRS | 5 years
  Self-reported substance use for youth as measured by the NM-YRRS
Feelings of safety measured by the NM-YRRS | 5 years
  Self-Reported experiences of bullying and safety concerns for youth as measured by the NM-YRRS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Willging CE, Green AE, Ramos MM. Implementing school nursing strategies to reduce LGBTQ adolescent suicide: a randomized cluster trial study protocol. Implement Sci. 2016 Oct 22;11(1):145. doi: 10.1186/s13012-016-0507-2. PMID 27770819